CLINICAL TRIAL: NCT06509347
Title: Stabilometry After Pressure Release of the Flexor Digitorum Brevis Muscle Versus a Non-emission Laser: Clinical Trial
Brief Title: Stabilometry After Pressure Release of the Flexor Digitorum Brevis Muscle Versus a Non-emission Laser.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayuben Private Clinic (Other)
Responsible Party: Principal Investigator, EVA MARIA MARTÍNEZ JIMENEZ, Physiotherapist responsible area, Mayuben Private Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1912202200923A
Record Dates: First submitted 2024-07-07; First posted 2024-07-19 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Balance; Manual Therapy; Foot; Myofascial Pain Syndrome; Myofascial Trigger Point
Keywords: balance; myofascial trigger point; foot
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant
Masking Description: Laser is a non-emission Laser
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pressure release (Experimental): Application of pressure on the trigger point of the flexor digitorum brevis until remission of referred pain for a minimum of 90 seconds, at least 3 cycles.
  Interventions: Other: Preassure release
- Non-emision Laser (Sham Comparator): Application of a non-emitting laser for 5 minutes on the trigger point of the flexor digitorum brevis muscle.
  Interventions: Other: Non-emision laser

INTERVENTIONS:
Other: Preassure release — Preassure release in Flexor digitorum brevis trigger point muscle.
  Arms: Pressure release
Other: Non-emision laser — Bilateral non emission Laser in latent trigger points of the Flexor digitorum Brevis Muscle
  Arms: Non-emision Laser

SUMMARY:
In this study we will test the effects of pressure release on the Flexor digitorum brevis muscle on stabilometric variables that support static equilibrium.

DETAILED DESCRIPTION:
In this study we will test the effects of pressure release on the Flexor digitorum brevis muscle on the stabilometric variables that support static balance. To test the effects on balance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Must have latent trigger point in Flexor Brevis Digitorum muscles with no other pathologies.

Exclusion Criteria:

* Previous lower extremities surgery.
* History of lower extremities injury with residual symptoms (pain, "giving-away" sensations) within the last year.
* Leg-length discrepancy more than 1 cm
* Balance deficits (determined by oral questionnaire regarding falls)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2024-07-22 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
1.Stabilometric variable x displacement open eyes before pressure release. | Through study completion, an average of 1 week.
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in X (in millimeters) with open eyes.
2.Stabilometric variable x displacement open eyes before non emission Laser | Through study completion, an average of 1 week.
  Stabilometry assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure displacement of the center of pressures in Y (in millimeters) with open eyes.
3.Stabilometric variable center of pressure area open eyes before pressure release. | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure displacement of the center of Pressure (COP) area (in millimeters²) with eyes open.
4.Stabilometric variable center of pressure area open eyes before non emission laser. | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure displacement of the center of Pressure (COP) area (in millimeters²) with eyes open.
5.Stabilometric variable center of pressure speed displacement of the anteroposterior(a-p) direction open eyes before pressure release. | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in millimeters/second).
6.Stabilometric variable center of pressure speed displacement of the anteroposterior(a-p) direction open eyes before pressure non-emission Laser. | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in millimeters/second).
7.Stabilometric variable y displacement open eyes before pressure release | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure displacement of the center of pressures in Y (in millimeters) with open eyes.
8.Stabilometric variable x displacement open eyes before non emission Laser | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure displacement of the center of pressures in Y (in millimeters) with open eyes.
9.Stabilometric variable center of pressure speed displacement of the latero-lateral(lat-lat) direction open eyes before pressure release | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in millimeters/second).
10.Stabilometric variable center of pressure speed displacement of the latero-lateral(lat-lat) direction open eyes non emision Laser. | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometry variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in millimeters/second).
11.Stabilometric variable x displacement closed eyes before pressure release | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure displacement of the center of pressures in X (in millimeters) with closed eyes.
12.Stabilometric variable x displacement closed eyes before non emission Laser | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure displacement of the center of pressures in X (in millimeters) with closed eyes.
13.Stabilometric variable center of pressure area closed eyes before pressure release. | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure displacement of the center of Pressure (COP) area (in millimeters²) with closed eyes.
14.Stabilometric variable center of pressure area closed eyes before non emission laser. | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure displacement of the center of Pressure (COP) area (in millimeters²) with closed eyes.
15.5.Stabilometric variable center of pressure speed displacement of the anteroposterior(a-p) direction closed eyes before pressure release. | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in millimeters/second).
.Stabilometric variable center of pressure speed displacement of the anteroposterior(a-p) direction closed eyes before pressure non-emission Laser. | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure center of pressure speed displacement of the anteroposterior(a-p) direction (in millimeters/second).
17.Stabilometric variable y displacement closed eyes before pressure release | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure displacement of the center of pressures in Y (in millimeters) with closed eyes.
18.Stabilometric variable x displacement closed eyes before non emission Laser | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure displacement of the center of pressures in Y (in millimeters) with closed eyes.
9.Stabilometric variable center of pressure speed displacement of the latero-lateral(lat-lat) direction closed eyes before pressure release. | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in millimeters/second).
20. Stabilometric variable center of pressure speed displacement of the latero-lateral(lat-lat) direction closed eyes non emission Laser. | Through study completion, an average of 1 week.
  Stabilometric assessment was used and subjects were instructed to stand barefoot on the force platform, participants were instructed to remain in a relaxed standing posture with feet shoulder-width apart and positioned at 30º away from the midline. Stabilometric variables measure center of pressure speed displacement of the latero-lateral(lat-lat) direction (in millimeters/second).

CONTACTS AND LOCATIONS:
Locations (1):
- Eva María Martínez-Jiménez In Mayuben CLinic, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martinez-Jimenez EM, Becerro-de-Bengoa-Vallejo R, Losa-Iglesias ME, Perez-Boal E, Posada-Ordax J, Sanchez-Serena A, Trevisson-Redondo B, Benito-de-Pedro M, Martinez-Corcoles V, Casado-Hernandez I. Plantar pressures and stabilometry effects of ischemic compression in Flexor digitorum brevis muscle Myofascial Trigger Point: A prepost study. PLoS One. 2025 Aug 14;20(8):e0329734. doi: 10.1371/journal.pone.0329734. eCollection 2025. PMID 40811690